CLINICAL TRIAL: NCT06444490
Title: Comparison of Oral Hygiene Instruction Methods on Oral Hygiene Behaviour Among Older Adults
Brief Title: Oral Hygiene Among Portuguese Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Egas Moniz - Cooperativa de Ensino Superior, CRL (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PHDICS
Record Dates: First submitted 2024-05-29; First posted 2024-06-05 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-05

CONDITIONS: Oral Hygiene; Oral Health; Older
Keywords: oral hygiene; oral health; health motivation; toothbrushing; dental devices; self-perception

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- General Approach (GA) (Active Comparator): This approach consisted of a 15-minute session in which the dentist attempted to impart knowledge about oral hygiene in general, highlighting some of the most common situations in this age group, namely the difficulty in achieving correct brushing and flossing, demonstrating the correct technique on a typodont (model), and alerting them to the importance of oral health to general health. Periodontal disease, tooth decay and denture care were also covered in general terms. Participants were given a written explanatory guide to reinforce good oral hygiene habits and an explanation of these diseases or conditions. Appropriate oral hygiene tools were also provided to encourage the expected improvement in oral health. Finally, there was a question-and-answer session to clarify any doubts the participant might have.
  Interventions: Behavioral: General Approach Instruction
- Personalised Technique (PT) (Active Comparator): This approach began with a self-examination in an extra-oral mirror by the participant to allow the professional to understand participant's perception of oral health, and the use of a plaque-disclosing solution to allow the participant to be more sensitive to the areas where brushing and flossing were not effective. Conditions such as caries lesions, major gingival recessions, areas of greater inflammation, areas where plaque accumulation or even tartar was more visible and further denture care were highlighted. The typodont (model) was then used to demonstrate the correct brushing and flossing technique. The session ended with the participant receiving an explanatory guide, a personalized plan, and more appropriate tools to promote the expected improvement in oral health. A question-and-answer session was used to clarify any doubts. This method took about approximately 20 minutes.
  Interventions: Behavioral: Personalised Technique Instruction

INTERVENTIONS:
Behavioral: General Approach Instruction — Oral health instruction focused more broadly on the different topics of oral diseases and oral hygiene care.
  Arms: General Approach (GA)
Behavioral: Personalised Technique Instruction — Oral health instruction based on the specific needs of each participant.
  Arms: Personalised Technique (PT)

SUMMARY:
The goal of this clinical trial was to compare two different oral hygiene instruction methods on oral hygiene behavior in older adults. We also wanted to evaluate the self-perception of oral health changes with each instruction method. The main questions we aim to answer were:

* Which method has better results in changing oral hygiene habits?
* Which method has better results in reducing bacterial plaque?

Participants:

* Completed a questionnaire about socioeconomic aspects and oral hygiene habits;
* Were examined to assess their oral hygiene status;
* Completed a questionnaire about self-perception of oral health;
* Received oral hygiene instruction (depending on the group: Generalised Approach or Personalised Technique).

Two months later, they were assessed again on oral hygiene habits, oral hygiene status, and self-perception of oral health.

DETAILED DESCRIPTION:
This study aimed to evaluate the effectiveness of two different oral hygiene instruction methods on oral hygiene behavior in older adults. Secondly, we intended to assess the self-perception of oral health changes with each instruction method.

This study was a clinical trial that included a convenience sample of 60 participants attending a university dental hospital (Egas Moniz Dental Clinic, Almada, Portugal).

Data were collected in two phases: The first phase (baseline) consisted of three parts: a questionnaire focusing on the participant's socioeconomic data and oral hygiene behaviors, clinical records obtained through an intraoral examination, using the Oral Hygiene Index-Simplified (OHI-S), and oral hygiene instruction.

For the oral hygiene instruction, the sample was divided into two groups of 30 participants (n=30) each group, exposed to different methods of professional education. The first one, identified as "General Approach" (GA), focuses more broadly on the different topics of oral diseases and oral hygiene care. The second group, identified as "Personalised Technique" (PT), was based on the specific needs of each participant.

After two months, to establish a follow-up session, the self-reported questionnaire on oral hygiene behavior and self-perceived oral health was administered again and the same clinical records on OHI-S were collected.

ELIGIBILITY:
Inclusion Criteria:

* Being able to speak and understand Portuguese;
* Being able to understand and sign an informed consent form;
* Being literate and able to comply with the study protocol.

Exclusion Criteria:

* Being edentulous;
* Being institutionalized;
* Having disabilities such as blindness, deafness, or dementia.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-01-30 (Actual); Primary Completion 2023-05-29 (Actual); Study Completion 2023-05-29 (Actual)

PRIMARY OUTCOMES:
Brushing frequency | 2 months
  Assessment of toothbrushing frequency (<2x/day or ≥ 2x/day)
Interdental devices usage | 2 months
  Assessment of dental floss or interdental brushes usage (yes/no)
Denture hygiene | 2 months
  Assessment of daily denture cleaning (yes/no)
Denture care | 2 months
  Assess whether participants sleep with their dentures in (yes/no)
Oral Hygiene Clinical Indicator | 2 months
  Assessment of Oral Hygiene Index - Simplified (OHI-S) (Greene & Vermillion, 1964). The six surfaces examined for the OHI-S are selected from four posterior and two anterior teeth. For posterior teeth, the buccal surfaces of the selected upper molars (usually 16 and 26) and the lingual surfaces of the selected lower molars (usually 36 or 46) are examined. For the incisors, the labial surfaces of the upper right central incisor (11) and the lower left central incisor (31) are evaluated.
  A score from 0 to 3 was then recorded for each surface, according to the classification for each index (debris or calculus). For each participant, the debris or calculus index was obtained by summing the scores and dividing by the number of surfaces scored.
  The Simplified Oral Hygiene Index is the sum of the Debris Index and the Calculus Index and can range from 0 to 6, with higher scores indicating poorer oral hygiene.
Treatment needs (oral clinical observation) | 2 months
  Assessment of participants' treatment needs (yes/no)

SECONDARY OUTCOMES:
Self-perception of oral health | 2 months
  Assess the participants' perception of oral health (poor/good)
Xerostomia | 2 months
  Assessment of dry mouth perception (yes/no)
Perceived treatment needs | 2 months
  Assessment of participants' perception of need for treatment (yes/no)

CONTACTS AND LOCATIONS:
Overall Officials: Inês C Santos, MSc, Principal Investigator — Egas Moniz School of Health & Science
Locations (1):
- Egas Moniz Dental Clinic, Almada, Caparica, Portugal

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie will result in a publication.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD will become available immediately after publication.
Access Criteria: Data will be available upon reasonable request. The Principal Investigator will review requests.

REFERENCES:
- [Background] GREENE JC, VERMILLION JR. THE SIMPLIFIED ORAL HYGIENE INDEX. J Am Dent Assoc. 1964 Jan;68:7-13. doi: 10.14219/jada.archive.1964.0034. No abstract available. PMID 14076341